CLINICAL TRIAL: NCT01102634
Title: Effects of Acu-Transcutaneous Electrical Nerve Stimulation (Acu-TENS) on Post-exercise Blood Lactate and Excessive Post-exercise Oxygen Consumption (EPOC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Prof. Alice Jones, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20100407006
Record Dates: First submitted 2010-04-08; First posted 2010-04-13 (Estimated); Last update posted 2010-04-13 (Estimated); Status verified 2010-04

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Acu-TENS (Experimental): Application of TENS over acupuncture points
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)
- Placebo-TENS (Placebo Comparator): Application of Acu-TENS but with no electricity
  Interventions: Device: Transcutaneous electrical nerve stimulation (TENS)

INTERVENTIONS:
Device: Transcutaneous electrical nerve stimulation (TENS) — Application of TENS over acupuncture points
  Arms: Acu-TENS
Device: Transcutaneous electrical nerve stimulation (TENS) — Placebo
  Arms: Placebo-TENS

SUMMARY:
The study aims to investigate the effect of Acu-TENS on post-exercise blood lactate level and EPOC

ELIGIBILITY:
Inclusion Criteria:

* with normal health (no known history of cardiovascular, pulmonary, metabolic or musculoskeletal diseases)

Exclusion Criteria:

* unable to communicate and follow the exercise procedures

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-04; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Blood lactate level | Before exercise
  Finger pick method - measured by Lactate Plus (Nova Biomedical, USA)
Blood lactate level | Immediately post exercise
  Finger pick method - measured by Lactate Plus (Nova Biomedical, USA)
Blood lactate level | 15 minutes post exercise
  Finger pick method - measured by Lactate Plus (Nova Biomedical, USA)
Oxygen consumption | Measurements continued during exercise and until heart rate returned to baseline
  measured by K4b2 (Cosmed, Italy)

SECONDARY OUTCOMES:
Heart rate | Measurements continued during exercise and until heart rate returned to baseline
  measured by Polar heart rate monitor (RS800CX, Polar Electro, Finland)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Jones, PhD, FACP, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Cardiopulmonary and Exercise Physiology Laboratory, The Hong Kong Polytechnic University, Hong Kong, Hong Kong, China